CLINICAL TRIAL: NCT02551991
Title: A Randomized, Open-label Phase 2 Study of Nanoliposomal Irinotecan (Nal-IRI)-Containing Regimens Versus Nab-Paclitaxel Plus Gemcitabine in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Study of Nanoliposomal Irinotecan (Nal-IRI)-Containing Regimens Versus Nab-paclitaxel Plus Gemcitabine in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-398-07-02-03; 2015-003086-28 (EudraCT Number)
Record Dates: First submitted 2015-09-10; First posted 2015-09-16 (Estimated); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; MM-398; Metastatic pancreatic cancer; First line pancreatic cancer treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nal-IRI + 5-FU/LV + oxaliplatin (Experimental)
  Interventions: Drug: nal-IRI; Drug: 5 fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: nal-IRI
  Other Names: MM-398
Drug: 5 fluorouracil
  Other Names: 5-FU
Drug: Leucovorin
  Other Names: LV
Drug: Oxaliplatin

SUMMARY:
This is an open-label, phase 2 non-comparative study to assess the safety, tolerability, and preliminary efficacy of nal-IRI in combination with other anticancer therapies in patients not previously treated for metastatic pancreatic adenocarcinoma. This study will assess the following regimen:

• nal-IRI + 5-fluorouracil (5-FU)/leucovorin (LV) + oxaliplatin

The study will be conducted in two parts:

Part 1, consisting of an initial dose exploration (Part 1A) followed by dose expansion (Part 1B) of the irinotecan liposome injection +5-FU/LV + oxaliplatin regimen and Part 2, consisting of a comparison of irinotecan liposome injection-containing regimen versus nab-paclitaxel plus gemcitabine. The comparative Part 2 was removed in a protocol amendment, dated 11 April 2018 (Version 6.0), before it was initiated, as this comparative part of the study is being undertaken as a stand-alone phase III study D-US-60010-001. This CSR only pertains to the single-arm dose exploration and dose expansion Part 1 results and no further reference is made to the comparative Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas that has not been previously treated in the metastatic setting
* Unresectable, locally advanced or metastatic disease; diagnosed within 6 weeks prior to screening
* At least one tumor lesion measurable by CT or MRI scan (according to RECIST v1.1)
* ECOG performance status of 0 or 1 at screening and within 72 hours prior to first dose if first dose occurs more than 72 hours post-screening
* Adequate hematological, hepatic, renal and cardiac function
* Recovered from the effects of any prior surgery or radiotherapy
* Patient has a Karnofsky performance status (KPS) ≥ 70 at Screening, and within 72 hours prior to date of first dose if first dose occurs more than 72 hours after screening (Part 1B only)

Exclusion Criteria:

* Prior treatment of pancreatic cancer in the metastatic setting (or locally advanced setting) with surgery (placement of stent is allowed), radiotherapy, chemotherapy or investigational therapy
* Prior treatment of pancreatic cancer with chemotherapy in adjuvant setting, except those where at least 12 months have elapsed since completion of the last dose and no persistent treatment-related toxicities present
* Uncontrolled Central Nervous System (CNS) metastases
* Clinically significant gastrointestinal disorder
* History of any second malignancy in the last 3 years. Patients with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible
* Presence of any contraindications for nal-IRI, irinotecan, 5-FU, leucovorin, oxaliplatin
* Use of strong CYP3A4 or inducers or presence of any other contra indications for irinotecan
* Pregnant or breast feeding
* Neuroendocrine or acinar pancreatic carcinoma
* Serum albumin < 3 g/dL at screening visit and within 72 hours prior to first dose if first dose occurs more than 72 hours post screening
* Patients with symptoms and signs of clinically unacceptable deterioration of primary disease at time of screening
* Previous treatment with irinotecan-based, nab-paclitaxel-based or gemcitabine-based resulting in disease progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (36):
- United States (29):
  - University of South Alabama, Mobile, Alabama
  - University of South Alabama - Mobile, Mobile, Alabama
  - Arizona Center for Cancer Care, Avondale, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UCLA Hematology Oncology - Ventura, Los Angeles, California
  - University of California Irvine Medical Center (UCIMC) - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado (CU) Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Eastern Maine Medical Cancer Care, Brewer, Maine
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Mayo Clinic Cancer Center - Rochester, Rochester, Minnesota
  - Oncology Hematology West PC dba Nebraska, Omaha, Nebraska
  - US Oncology - Comprehensive Cancer Centers of Nevada (CCCN), Las Vegas, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Oncology/Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center (OUHSC) Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute & Research Center, Eugene, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Medical Group of the Carolinas - Spartanburg Regional Health Services, Spartanburg, South Carolina
  - Texas Oncology Methodist Dallas Cancer Center, Dallas, Texas
  - Texas Oncology-Fort Worth 12 Ave, Fort Worth, Texas
  - Houston Methodist Cancer Center and Institute of Academic Medicine, Houston, Texas
  - Oncology Consultants - Houston, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center - Lubbock, Lubbock, Texas
  - Texas Oncology, P.A., San Antonio, Texas
- Australia (3):
  - St. John of God Health Care - Subiaco, Subiaco, Western Australia
  - Flinders Medical Centre, Bedford Park
  - Box Hill Hospital, Lilydale
- Spain (4):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Madrid Sanchinarro Centro Integral Oncologico Clara Campal (CIOCC), Madrid

REFERENCES:
- [Derived] Brendel K, Bekaii-Saab T, Boland PM, Dayyani F, Dean A, Macarulla T, Maxwell F, Mody K, Pedret-Dunn A, Wainberg ZA, Zhang B. Population pharmacokinetics of liposomal irinotecan in patients with cancer and exposure-safety analyses in patients with metastatic pancreatic cancer. CPT Pharmacometrics Syst Pharmacol. 2021 Dec;10(12):1550-1563. doi: 10.1002/psp4.12725. Epub 2021 Nov 20. PMID 34750990
- [Derived] Wainberg ZA, Bekaii-Saab T, Boland PM, Dayyani F, Macarulla T, Mody K, Belanger B, Maxwell F, Moore Y, Thiagalingam A, Wang T, Zhang B, Dean A. First-line liposomal irinotecan with oxaliplatin, 5-fluorouracil and leucovorin (NALIRIFOX) in pancreatic ductal adenocarcinoma: A phase I/II study. Eur J Cancer. 2021 Jul;151:14-24. doi: 10.1016/j.ejca.2021.03.028. Epub 2021 May 4. PMID 33957442
- [Derived] Liu X, Jiang J, Chan R, Ji Y, Lu J, Liao YP, Okene M, Lin J, Lin P, Chang CH, Wang X, Tang I, Zheng E, Qiu W, Wainberg ZA, Nel AE, Meng H. Improved Efficacy and Reduced Toxicity Using a Custom-Designed Irinotecan-Delivering Silicasome for Orthotopic Colon Cancer. ACS Nano. 2019 Jan 22;13(1):38-53. doi: 10.1021/acsnano.8b06164. Epub 2018 Dec 11. PMID 30525443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2 non-comparative, open-label study was conducted in previously untreated metastatic pancreatic cancer participants at 15 investigational sites in Australia, Spain and USA between 19 October 2015 and 15 February 2021.
Pre-assignment Details: This study was divided into 2 parts: Part 1 (dose exploration [Part 1A] followed by dose expansion [Part 1B] of the irinotecan liposome injection + 5 fluorouracil [5-FU]/leucovorin [LV] + oxaliplatin regimen) and Part 2 (comparison of irinotecan liposome injection-containing regimen versus [vs] nab-paclitaxel plus gemcitabine). Overall, 56 participants were enrolled in this study.
Groups:
- Dose Exploration: Cohort 1: Participants received irinotecan liposome injection 70 milligram per square meter (mg/m^2) followed by oxaliplatin 60 mg/m^2 followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Dose Exploration: Cohort -1; Dose Expansion: Cohort -1: Participants received irinotecan liposome injection 50 mg/m^2 followed by oxaliplatin 60 mg/m^2 followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 IV infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Dose Exploration: Cohort -2B: Participants received irinotecan liposome injection 50 mg/m^2 followed by oxaliplatin 85 mg/m^2 followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 IV infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Dose Exploration: Cohort -3: Participants received irinotecan liposome injection 55 mg/m^2 followed by oxaliplatin 70 mg/m^2 followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 IV infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1
Started | 7 | 7 | 10 | 7 | 25
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 10 | 7 | 25
Not completed — Death | 5 | 7 | 8 | 7 | 17
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 1 | 0 | 5
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least 1 dose of any study treatment.
Groups:
- Dose Exploration: Cohort 1: Participants received irinotecan liposome injection 70 mg/m^2 followed by oxaliplatin 60 mg/m^2 followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 IV infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Total
Number analyzed (Participants) | 7 | 7 | 10 | 7 | 25 | 56
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 4 | 4 | 3 | 4 | 19 | 34
  >= 65 years | 3 | 3 | 7 | 3 | 6 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 2 | 14 | 28
  Male | 1 | 3 | 8 | 5 | 11 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 7 | 9 | 7 | 21 | 50
  Black or African American | 0 | 0 | 0 | 0 | 2 | 2
  Asian | 1 | 0 | 1 | 0 | 1 | 3
  Not Reportable | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 7 | 7 | 10 | 7 | 21 | 52

OUTCOME MEASURES:

1. Primary Outcome: Part 1A: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: Adverse events (AEs) were considered to be DLTs if they occurred during the safety evaluation period (i.e, 28 days of Cycle 1; or 14 days after the second dose of study treatment if there was a treatment delay) and were deemed related to the study treatment regimen. Any AE that was related to disease progression was not considered a DLT.
Time Frame: From the start of the first study treatment (Cycle 1 Day 1) up to 14 days after the second dose of study treatment, maximum of 42 days
Population: Safety population included participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3
Number analyzed (Participants) | 7 | 7 | 10 | 7
Participants | 2 | 1 | 2 | 0

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: The PFS was defined as the time from date of first study treatment to the first documented radiographical progression of disease (PD), per investigator using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, or death from any cause, whichever comes first. The PFS was calculated using Kaplan-Meier technique.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study treatment), every 8 weeks after first dose, end of treatment (EoT) visit, then every 2 months thereafter (maximum of 278 weeks).
Population: Safety population included participants who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort -1: Pooled: Participants received irinotecan liposome injection 50 mg/m^2 followed by oxaliplatin 60 mg/m^2 followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 IV infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Cohort -1: Pooled
Number analyzed (Participants) | 7 | 7 | 10 | 7 | 25 | 32
months | 9.7 [2.96 to NA] — Upper limit of confidence interval was not evaluable due to below the level of detection. | 32.3 [0.53 to NA] — Upper limit of confidence interval was not evaluable due to below the level of detection. | 9.2 [0.46 to NA] — Upper limit of confidence interval was not evaluable due to below the level of detection. | 3.8 [1.22 to 5.78] | 9.2 [7.59 to 11.20] | 9.2 [7.59 to 11.96]

3. Secondary Outcome: Best Overall Response (BOR)
Description: The BOR was defined as the best response (complete response [CR] + partial response [PR] + stable disease [SD]) recorded from the start of study treatment until disease progression or start of new anticancer therapy using RECIST Version 1.1.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study treatment), every 8 weeks after first dose, EoT visit, then every 2 months thereafter (maximum of 278 weeks).
Population: Safety population included participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Cohort -1: Pooled
Number analyzed (Participants) | 7 | 7 | 10 | 7 | 25 | 32
Participants | 2 | 6 | 4 | 4 | 20 | 26

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with a BOR characterized as either a CR or PR relative to the total number of evaluable participants using RECIST Version 1.1. Evaluable participants were defined as treated participants with measurable disease at baseline.
Time Frame: as for outcome 3
Population: Safety population included participants who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Cohort -1: Pooled
Number analyzed (Participants) | 7 | 7 | 10 | 7 | 25 | 32
percentage of participants | 0 [0 to 41.0] | 42.9 [9.9 to 81.6] | 30.0 [6.7 to 65.2] | 14.3 [0.4 to 57.9] | 32.0 [14.9 to 53.5] | 34.4 [18.6 to 53.2]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as percentage of participants with CR or PR or SD or Non-PD/Non-CR, per RECIST Version 1.1 relative to total number of treated participants with measurable disease at baseline.
Time Frame: At Week 16
Population: Safety population included participants who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Cohort -1: Pooled
Number analyzed (Participants) | 7 | 7 | 10 | 7 | 25 | 32
percentage of participants | 42.9 [9.9 to 81.6] | 71.4 [29.0 to 96.3] | 40.0 [12.2 to 73.8] | 28.6 [3.7 to 71.0] | 72.0 [50.6 to 87.9] | 71.9 [53.3 to 86.3]

6. Secondary Outcome: Median Overall Survival (OS)
Description: The OS was the time from date of first study treatment to the date of death from any cause. Participant survival data were collected from all available sources. The OS was calculated using Kaplan-Meier technique.
Time Frame: as for outcome 3
Population: Safety population included participants who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Cohort -1: Pooled
Number analyzed (Participants) | 7 | 7 | 10 | 7 | 25 | 32
months | 12.6 [3.98 to 21.03] | 12.5 [0.53 to 12.71] | 16.6 [0.69 to 26.74] | 5.8 [1.35 to 14.65] | 12.7 [8.18 to 23.66] | 12.6 [8.74 to 19.12]

7. Secondary Outcome: Median Duration of Response (DoR)
Description: The DoR was defined as the time from the first date of response (CR or PR) to first date of documented radiographical PD, per investigator using RECIST Version 1.1. This only applied to participants with CR or PR. If a participant was given a new anticancer therapy prior to first response, DoR was not calculated. The DoR was calculated using Kaplan-Meier technique.
Time Frame: as for outcome 3
Population: Safety population included participants who received at least 1 dose of any study treatment. Only participants with DoR events were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1 | Cohort -1: Pooled
Number analyzed (Participants) | 0 | 2 | 1 | 0 | 4 | 6
months |  | 28.4 [3.52 to NA] — Upper limit of confidence interval was not evaluable due to below the level of detection. | NA [NA to 16.39] — Median and lower limit of confidence interval was not evaluable due to below the level of detection. |  | 9.4 [2.20 to NA] — Upper limit of confidence interval was not evaluable due to below the level of detection. | 9.4 [3.52 to NA] — Upper limit of confidence interval was not evaluable due to below the level of detection.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported from the time of first study treatment administration (Day 1) up to 30 days after the date of last study treatment administration or until the start of alternative anticancer therapy, approximately 1008 days. All-Cause Mortality are reported from first participant enrolled to last participant died, approximately 1946 days.
Description: Safety population included participants who received at least 1 dose of any study treatment.
Arm/Group | Dose Exploration: Cohort 1 | Dose Exploration: Cohort -1 | Dose Exploration: Cohort -2B | Dose Exploration: Cohort -3 | Dose Expansion: Cohort -1
All-Cause Mortality (participants affected / at risk) | 5/7 | 7/7 | 8/10 | 7/7 | 17/25
Serious Adverse Events (participants affected / at risk) | 6/7 | 2/7 | 7/10 | 4/7 | 15/25
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 10/10 | 7/7 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Exploration: Cohort 1 (N=7) | Dose Exploration: Cohort -1 (N=7) | Dose Exploration: Cohort -2B (N=10) | Dose Exploration: Cohort -3 (N=7) | Dose Expansion: Cohort -1 (N=25)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Anaemia of Malignant Disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary Dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriospasm Coronary (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Exploration: Cohort 1 (N=7) | Dose Exploration: Cohort -1 (N=7) | Dose Exploration: Cohort -2B (N=10) | Dose Exploration: Cohort -3 (N=7) | Dose Expansion: Cohort -1 (N=25)
Nausea (Gastrointestinal disorders) | 5 (9) | 6 (7) | 9 (19) | 5 (6) | 23 (49)
Diarrhoea (Gastrointestinal disorders) | 6 (18) | 5 (22) | 6 (14) | 6 (14) | 22 (54)
Vomiting (Gastrointestinal disorders) | 5 (12) | 4 (7) | 5 (8) | 3 (4) | 14 (28)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (9) | 4 (5) | 1 (2) | 13 (22)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 3 (5) | 3 (3) | 4 (6) | 8 (16)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (7) | 1 (1) | 7 (9)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (9) | 5 (10) | 7 (13) | 5 (6) | 16 (21)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 5 (14)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (15)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 1 (3) | 1 (1) | 2 (2)
Chills (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (10) | 6 (9) | 4 (8) | 3 (4) | 12 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (3) | 5 (6) | 3 (11) | 12 (34)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 3 (3) | 3 (4) | 2 (2) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 2 (3) | 2 (2) | 4 (21)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 2 (3) | 1 (1) | 3 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (18)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (18)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (5) | 2 (2) | 3 (6) | 2 (2) | 8 (9)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 3 (6) | 2 (3) | 2 (5) | 7 (11)
Dysgeusia (Nervous system disorders) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 4 (5)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 3 (5) | 0 (0) | 2 (7)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lhermitte's sign (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 3 (13) | 5 (6) | 1 (2) | 10 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (10) | 4 (4) | 0 (0) | 9 (18)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 3 (5) | 2 (2) | 7 (35)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 2 (3) | 4 (6) | 2 (4) | 5 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (17)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 9 (15)
Platelet count decreased (Investigations) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 5 (17)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (10)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (7) | 1 (1) | 4 (12)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (17)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (23)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung diffusion test decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 5 (6) | 1 (1) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (5) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The comparative Part 2 was removed in a protocol amendment, dated 11 April 2018, before it was initiated, as this comparative part of the study is being undertaken as a stand-alone Phase 3 study D-US-60010-001.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT02551991/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02551991/SAP_001.pdf